CLINICAL TRIAL: NCT04583059
Title: Effect of Ankle Taping and Bandaging on Balance and Proprioception Among Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Gelisim University (Other)
Responsible Party: Principal Investigator, Motaz Alawna, Assistant Professor (Principal Investigator), Istanbul Gelisim University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Taping, Bandaging
Record Dates: First submitted 2020-10-04; First posted 2020-10-12 (Actual); Last update posted 2020-10-12 (Actual); Status verified 2020-10

CONDITIONS: Ankle Injuries
MeSH Terms: conditions — Ankle Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Taping Group (Experimental): A hard-preventive Zinc oxide tape was used in this study. Taping procedure consists of three separate steps: First step involved application of the anchor tape, which achieved by applying the tape circumferentially just above the malleolar level at the lower end of the shank. Second step involved application of the stirrup. During this step, the foot was held in neutral, and the tape applied to pass from the medial side of the ankle, under the foot just over the heel area (posterior one-third of the foot) and up along the lateral side of the ankle. The second step was repeated to apply the second stirrup. Both ends of the stirrups were firmly attached to the anchor tape applied during the first step and this attachment was reinforced with a locking tape during the third and final step by once again applying the tape circumferentially just above the malleolar level at the lower end of the shank. Taping was applied by a physical therapist according to the health association requirements
  Interventions: Other: Taping
- Bandaging Group (Experimental): Standard 10 cm width elastic bandage was used. The elastic bandage was wrapped around the ankle joint to form an 8-figure shape starting from the forefoot. Then, the bandage was taken diagonally upwards, steeply enough to go well above the heel. Then, the bandage was taken around the lower calf area to form an anchor. Then its diagonally taken down across the midfoot. Again the bandage was wrapped around the forefoot and going diagonally up to finish off around the lower calf, leaving the heel open. During the bandage application process, the therapiest didn't stretch the bandage, because bandage does note need to be stretched during the application, as the bandage becomes naturally tight when its layers wraped over each others. the participant was asked to wear his/her sport shoes over the bandage during the measurement procedures.
  Interventions: Other: Taping

INTERVENTIONS:
Other: Taping — A hard-preventive Zinc oxide tape was used in this study. Taping procedure consists of three separate steps: First step involved application of the anchor tape, which achieved by applying the tape circumferentially just above the malleolar level at the lo

SUMMARY:
Leg length was measured (right and left leg) while the participant lying supine, from the anterior superior iliac spine to the inferior border of the ipsilateral medial malleoli by using standard measure tape. The dominant leg was determined according to Vauhnik. & ark. modified version. The limb that was used in at least 2 of the 3 following activities: (1). Kicking a ball, (2). Drawing a diamond figure on the ground and (3).using his leg and step over a spider toy was considered as the dominant leg.30

DETAILED DESCRIPTION:
Participants

Seventy-four healthy subjects participated in this study (37 male and 37 female). Healthy subjects were selected because ankle injuries frequently occur during normal locomotion; and most people, not only athletes, experience an ankle injury at least once during their entire life.25,27

Before starting this study power test was performed to determine the number of participants. Participant's age range was 18 - 30 years old and participants were recruited from university population, Participants were divided randomly into two groups (Taping group n=37) and (Bandaging group n=37. Participant were excluded if he/she reports (a) previous hip/pelvis, knee, ankle, or foot surgery within the past year; (b) lower extremity amputation; (c) injury to the lower extremities six months; (d) known balance impairment due to neurological disorder, vestibular disorder, medication use, or other; (f) pregnancy; or (g) concussion within the previous three months. Standard clinical stability testing of the ankle ligamentous structures was performed to rule out anterior and lateral talocrural joint instability and lower extremity injuries during the previous 6 months. Each volunteer signed an informed consent form before participation. This study was approved by Dokuz E|ylul university ethics committee.

Procedures Leg length was measured (right and left leg) while participant lying supine, from the anterior superior iliac spine to the inferior border of the ipsilateral medial malleoli by using standard measure tape. The dominant leg was determined according to Vauhnik. & ark. modified version. The limb that was used in at least 2 of the 3 following activities: (1). Kicking a ball, (2). Drawing a diamond figure on the ground and (3).using his leg and step over a spider toy, was considered as the dominant leg.30

Ankle taping Procedures Zinc oxide tape has been was used, its hard - preventive tap. The taping procedure consists of three separate steps: The first step involved the application of the anchor tape, which achieved by applying the tape circumferentially just above the malleolar level at the lower end of the shank. The second step involved the application of the stirrup. During this step, the foot was held in neutral, and the tape applied to pass from the medial side of the ankle, under the foot just over the heel area (posterior one-third of the foot) and up along the lateral side of the ankle. The second step was repeated to apply the second stirrup. Both ends of the stirrups were firmly attached to the anchor tape applied during the first step and this attachment was reinforced with a locking tape during the third and final step by once again applying the tape circumferentially just above the malleolar level at the lower end of the shank. The taping was applied by a physical therapist according to the health association requirements.23

Ankle bandaging Procedures Standard 10 cm width elastic bandage was used. The elastic bandage was wrapped around the ankle joint to form an 8-figure shape starting from the forefoot. Then the bandage is taken diagonally upwards, steeply enough to go well above the heel, then around the lower calf area to form an anchor, then diagonally down across the midfoot, again wrapped around the forefoot and going diagonally up to finish off around the lower calf, leaving the heel open.9 Then the participant was allowed to wear his/her sport shoes over the bandage during the measurement procedures.

Balance measurement Procedures Star Excursion Balance Test (SEBT) is a field test and widely used to assess dynamic postural control, and has an excellent interrater reliability (ICC = 0.86 - 0.92)12. In thıs study the SEBT was used to evaluate balance. 8 strips of athletic tape with a length of 6 feet were used. Then a '+' sign was formed. Then 'x' sign was formed with the other two strips. The lines were separated from each other by an angle of 45°. The participant was asked to wear sports clothes and take off the shoes, then to step on the center of the grid formed by eight lines using the dominant leg, the plantar aspect of the first metatarsophalangeal joint (ball of the foot) was positioned on the intersecting lines at the center of the grid to maintain consistency in foot placement. The participant starts to reach as possible as far in the eight lines, make a light touch on the line, and return the reaching leg back to the center, while maintaining a single-leg stance with the other leg in the center of the grid, starting from anterior direction and progressing clockwise. The order of the directional reaches was as follows: A, AM, M, PM, P, PL, L, AL. When reaching in the lateral and posterolateral directions, participants must reach behind the stance leg to complete the task.13

The participant practiced 6 training attempts to reduce the learning effect, and then after 5-min of rest period participant performed 3 trials in each of the 8 directions, 5-min of rest period was taken between each one of the three trials. The researcher recorded the reaching distance using standard tape measure by marking the tape as the distance from the center of the gird to the maximal reaching point, the average of these three attempts was calculated and then normalized to the leg length, the obtained result used in the statistical analysis. If the participant used the stance leg for a high amount of support, was unable to maintain balance on the stance leg, or removing his feet from the center any time while doing the trial, the attempt was canceled and repeated again. In the case of a rejected trial, verbal feedback was given to the participants so they attempt to correct the performance error(s) on the next trial.13

The balance measurements were done 4 times, (before ankle taping, after 20 minutes while using ankle taping, after 24 hours while using ankle taping and immediately after removing the tap (after 24 hours).

Proprioception measurement Procedures Invistigators used the measurement procedure which described in the study which was doneIris et al23. by The first step: volunteers were seated in a high chair, and while their eyes are closed, the researcher consecutively on different graduated surfaces (10° dorsiflexion, neutral position, 10° plantarflexion, and 20° plantarflexion) respectively, each position will be done for just one time and will be held for 5 seconds. The researcher told the volunteers that they have to memorize the positions because they have to do it again by themselves. Simultaneously, each joint position was recorded to obtain the target angle using the universal goniometer. This was the angle that the volunteer was instructed to reproduce during the testing part of the study. The second step: The volunteer was then encouraged to walk freely next to the researcher for 10 minutes, still blindfolded. The third step: Then the volunteer sat on a high chair that did not allow his or her feet to touch the floor (to avoid any information from the sole). Finally, the researcher encouraged the subject to reproduce the four memorized positions, starting from and finishing in the neutral position each time. The volunteer maintained each ankle position, announced by the researcher at random, for five seconds. The volunteer's ankle movement was recorded using the universal goniometer, and this reproduced ankle angle was called the estimated angle.

The difference between the learned positions and the positions that were done by the volunteer was calculated and documented. Deviation from the learned angle (degrees) described the direction of Error when subjects tried to reproduce the requested position. Deviation was obtained by coding net Error, which was based on the correct position occurring when the learned and estimated angle were equal (±5 degrees)23.

The position (ROM) measurements were done on four occasions, (before ankle external support, after 20 minutes while using external support, after 24 hours while using external support and immediately after removing the external support (after 24 hours).

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Non-athletes

Exclusion Criteria:

* Previous hip/pelvis, knee, ankle, or foot surgery within the past year
* Lower extremity amputation
* Injury to the lower extremities six months
* Known balance impairment due to neurological disorder, vestibular disorder, medication use, or other
* Pregnancy
* Concussion within the previous three months

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 74 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Balance | 2 Months
  Star Excursion Balance Test used to evaluate balance. Participant was asked to wear sport without shoes, then to step on the center of the grid by the dominant leg, plantar aspect of the first metatarsophalangeal joint was positioned at the center of the grid. Participant starts reaching as possible as far in the eight lines, make a light touch on the line, and return reaching leg back to center, while maintaining a single-leg stance with other leg at the grid center, starting from anterior direction, progressing clockwise. The order of the reaches as follows: A (anterior), AM (anteromedial), M (medial), PM (posteromedial), P (posterior), PL (posterolateral), L (lateral), AL (anterolateral). During the lateral and posterolateral directions, participants must reach behind the stance leg to complete task. These measurements were done 4 times, (before ankle taping, after 20 minutes while using ankle taping, after 24 hours while using ankle taping and immediately after removing the tap
Proprioception | 2 Months
  First step: volunteers seated in a high chair, while their eyes are closed, the researcher consecutively on different graduated surfaces (10° dorsiflexion, neutral position, 10° plantarflexion, 20° plantarflexion) each position was done for one time and held for 5 seconds. Researcher told volunteers that they have to memorize the positions to do it again themselves. Each position recorded to obtain the target angle using the universal goniometer. Second step: Volunteer encouraged to walk freely next to the researcher for 10 minutes, still blindfolded. Third step: volunteer sat on a high chair that did not allow his or her feet to touch the floor. Finally, the researcher encouraged the subject to reproduce the four memorized positions. Volunteer maintained each ankle position, announced by the researcher at random, for five seconds. These measurement were done four times (before, after 20 minutes, after 24 hours of using external support and immediately after removing external support

CONTACTS AND LOCATIONS:
Locations (1):
- Motaz Alawna, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No